CLINICAL TRIAL: NCT01912430
Title: Retrospective Data Analysis of the Impact of Vital Care Targeted Population Management Upon a Matched Cohort of Scott and White Health Plan Beneficiaries
Brief Title: Retrospective Data Analysis of VitalCare Targeted Population Management on Scott and White Chronically Ill Beneficiaries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scott & White Health Plan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 120246
Record Dates: First submitted 2013-07-18; First posted 2013-07-31 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: Chronic Illness
Keywords: Integrated Care Coaching; Chronic Care Coaching; Care Coaching
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ICC (Integrated Care Coaching) (Experimental): Received evidence-based, protocol-driven integrated care coaching intervention to improve chronic illness health outcomes (clinical, financial).
  Interventions: Behavioral: ICC (Integrated Care Coaching) Intervention Group
- Control Group (Experimental): Matched cohort by age and chronic illness diagnoses - no intervention
  Interventions: Behavioral: ICC (Integrated Care Coaching) Intervention Group

INTERVENTIONS:
Behavioral: ICC (Integrated Care Coaching) Intervention Group
  Other Names: Health Integrated Inc. Integrated Care Coaching (ICC)

SUMMARY:
New payment methods such as Accountable Care Organization (ACO's) and medical homes facilitate are new models for providers to deliver cost effective, quality patient outcomes. Integrated Care Coaching (ICC) is a healthcare delivery model combining telephonic interventions with an intelligent information technology platform that offered validated protocols and patient outcomes tracking. Health Integrated, Inc. has developed a validated program of Integrated Care Coaching (ICC), which was branded as "VitalCare", and implemented with over 7,000 members of the Scott and White Health Plan in Texas, would reduce healthcare costs/achieve a return on investment (ROI), improve clinical outcomes, and be satisfying for participants.

DETAILED DESCRIPTION:
A prospective, pre-post historical control design trial with a concurrent control group cost/satisfaction analysis with a retrospective clinical study was undertaken with adult, Scott and White Health Plan (SWHP) patients with chronic illnesses. From 2007 to 2010, a total of 7,411 ICC and 10,148 control patients participated. Variables were costs, return on investment (ROI), iterative Patient Health Questionnaire (PHQ)9 scores, and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Having one or more of 21 chronic conditions, including those with depression and multiple chronic comorbidities.

Exclusion Criteria:

* Presence of Major Cancer, HIV, or ESRD in either the baseline or measurement periods
* Claims in excess of $100,000 in either baseline or intervention period.
* Claims for long term care or hospice in either baseline or intervention period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17559 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Return of Investment and Cost of Medical Care | 6 to 12 months
  Primary outcomes were ROI and cost of medical care (including inpatient, outpatient, emergency room, office and other (ie, physical therapy). ICC participants and control group members had a minimum of 6 months to a maximum of 12 months measurement period.

SECONDARY OUTCOMES:
Level of Depressive Symptoms per Interactive Patient Health Questionnaire (PHQ-9) scores | 6 to 12 months
  Secondary outcome was level of depressive symptoms per Interactive Patient Health Questionnaire (PHQ-9) scores. ICC participants and control group members had a minimum of 6 months to a maximum of 12 months measurement period.

OTHER OUTCOMES:
Patient Satisfaction | 6 to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marylou Buyse, M.D., M.S., Principal Investigator — Scott and White Health Plan
Locations (1):
- Scott & White Health Plan, Temple, Texas, United States